CLINICAL TRIAL: NCT04318912
Title: An Observational Registry Study for Management of COPD Patients in China
Brief Title: An Observational Registry of Chinese COPD Study
Acronym: ORCHIDS
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongtao Niu, Resident Doctor, China-Japan Friendship Hospital
Other Study IDs: 21971
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: COPD
Keywords: COPD; health policy; telimedicine; management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: Adults age 40 or older with a diagnosis of chronic obstructive pulmonary disease (COPD) having been prescribed any COPD treatment (initial or subsequent) outside of a clinical trial.

SUMMARY:
This is a multi-center, observational registry study involving secondary and tertiary hospitals across China. The objective is to study the disease burden, disease progression, comorbidities, treatment pattern and real-world cost, effectiveness and safety of different therapy options for COPD patients in Chinese clinical practice in China.

DETAILED DESCRIPTION:
COPD is the most common chronic respiratory disease in China and has caused significant economic and humanistic burden. Patient reported outcomes (PRO) have been widely used to assess disease activity and quality of life for COPD patients. Wearable devices enable recording activity data of patients continuously and automatically. The objective of the study is to study the disease burden, disease progression, comorbidities, treatment pattern and real-world cost, effectiveness and safety of different therapy options for COPD patients in Chinese clinical practice in China. This is a multi-center, observational registry study involving secondary and tertiary hospitals across China. 3000-5000 participants are planned to be recruited. Each participant will be followed-up at baseline and every 3 months. Clinical assessment data, laboratory examination data and cost data are captured from electronic medical records (EMR). Patient-reported outcome (PRO) data are collected via smartphone app. Part of patients will receive wearable devices to record digital health technology (DHT) data. As the first ever observational registry focused on COPD stable-period management, this study can provide more information on these following issues. (1) Annual changes in COPD prevalence, treatment pattern and economic burden in China. (2) Assessing the real-world effectiveness and safety of different treatment patterns of COPD via EMR, PRO and DHT. (3) Cost-effectiveness and budget impact to the public healthcare funds of different treatment patterns of COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 40 or older with a diagnosis of chronic obstructive pulmonary disease (COPD) having been prescribed any COPD treatment (initial or subsequent) outside of a clinical trial.
2. Have plans for future visits at the site for continued management of COPD.

Exclusion Criteria:

1. Inability to provide written informed consent/assent.
2. Being enrolled in any interventional study or trial for COPD treatment. Note: Patient may be enrolled in other registries or studies where COPD treatment outcomes are observed and/or reported (such as center-based registries).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults age 40 or older with COPD having been prescribed any COPD treatment outside of a clinical trial. 3000-5000 patients are planned to be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Characterize COPD Disease Severity in Clinical Practice | 2 years
  Pulmonary Function Test measured by protable spirometer can represent the severity stages of COPD
Characterize COPD Disease Activity in Clinical Practice | 2 years
  Acute exacerbation of symptoms can reflect the disease activity and disease control of COPD.

SECONDARY OUTCOMES:
Evaluate Medical Expenditure in Clinical Practice | 2 years
  Medical expenditure for patients include inpatient cost, outpatient cost and emergency room cost.
Evaluate Patient Reported Outcome | 2 years
  COPD Assessment Test (CAT) is an 8-item, self-reported scale which can represent symptom and health status for COPD patients.
Evaluate Health Related Quality of Life | 2 years
  Euroqol-5 Dimension Questionnaire (EQ-5D) is an 5-item, self-reported scale which can measure health related quality of life.
Evaluate Digital Health Technology Outcome | 2 years
  Real-time monitoring of oxygen saturation (SpO2) is an objective manifestation of dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Study Director — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang X, Pan J, Fang F, Li Y, Lei J, Niu H, Li W, Dong F, Zheng Z, Peng Y, Yang T, Wang C, Jia C, Huang K. Characteristics and risk factors of patients with undiagnosed COPD in China: results of a nationwide study from the 'Happy Breathing' Programme with mixed methods evaluation. BMJ Health Care Inform. 2025 Oct 7;32(1):e101323. doi: 10.1136/bmjhci-2024-101323. PMID 41057271
- [Derived] Jia C, Zhang C, Fang F, Huang K, Dong F, Gu X, Niu H, Li S, Wang C, Yang T. Enjoying Breathing Program: A National Prospective Study Protocol to Improve Chronic Obstructive Pulmonary Disease Management in Chinese Primary Health Care. Int J Chron Obstruct Pulmon Dis. 2020 Sep 15;15:2179-2187. doi: 10.2147/COPD.S258479. eCollection 2020. PMID 32982210